CLINICAL TRIAL: NCT06495983
Title: Dynamic Hormone Profiling and Multimodal Data Capture in Primary Aldosteronism
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: REK 729178
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Mineralocorticoid Excess; Primary Aldosteronism; Hypercortisolism
Keywords: aldosterone
MeSH Terms: conditions — Hyperaldosteronism; Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — data from microdialysis fluid, blood and urine will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary aldosteronism: Patients with suspected and/or confirmed primary aldosteronism, aged 18-70 years
  Interventions: Device: dynamic microdialysis sampling

INTERVENTIONS:
Device: dynamic microdialysis sampling — Included patients will perform 24-hour dynamic microdialysis sampling from subcutaneous tissue fluid of the lower abdomen, applying the U-Rhythm sampler. Simutaneous measurements of blood pressure, glucose, and registration of activity level, meals and sleep pattern during microdialysis sampling may be performed. Microdialysis sampling will be performed during various conditions: during daily life activities, during saline infusion suppression testing and during dexamethasone suppression testing. Repeated sampling may be performed post treatment.

SUMMARY:
This study is a observational study applying 24-hour microdialysis methodology to perform dynamic multisteroid adrenal hormone profiling of patients with suspected or confirmed PA. Simultaneous registration of blood pressure, tissue glucose, sleep pattern, activity level and food intake registration may be performed. The overall objective is to develop a novel, sensitive, fast and user-friendly diagnostic procedure for PA, using multimodal data capture including dynamic multisteroid hormone profiling from microdialysis fluid.

DETAILED DESCRIPTION:
Primary aldosteronism is the most common cause of secondary hypertension. Primary aldosteronism has increased risk of organ complications compared with primary hypertension if left undiagnosed and without specific treatment. However, the current diagnostic work-up is a cumbersome, multistep process, relying on repeated single time point measurements of aldosterone, not capturing the rhythmic nature of aldosterone and related adrenal hormone secretion.

In this study we will apply the U-Rhythm microdialysis sampling system for 24-hour measurements from subcutaneous microdialysis fluid, analysed with LC/MS-MS methodology for dynamic multisteroid adrenal hormone profiling. We will further compare multisteroid hormone profiling results with variations in blood pressure and tissue glucose, sleep pattern, activity level and food intake.

The overall objective of the study is to develop a novel, sensitive, fast and user-friendly diagnostic procedure for PA, using multimodal data capture including 24-hour dynamic multisteroid hormone profiling from microdialysis tissue.

Primary objective

• Assess dynamic multisteroid rhythmicity in microdialysis fluid of aldosterone, precursors and metabolites of the mineralocorticoid and glucocorticoid pathway, compared to standard diagnostic work-up in patients with suspected or confirmed PA.

Secondary objectives

* Quantify the influence of salt and volume loading during diagnostic saline infusion test on multisteroid adrenal rhythmicity.
* Quantify the influence of glucocorticoids/ACTH suppression on multisteroid rhythmicity.
* Quantify the influence of cortisol co-secretion on multisteroid rhythmicity in PA.
* Quantify influence of blood pressure, pulse, sleep, food intake and movement on multisteroid rhythmicity in PA.

ELIGIBILITY:
Inclusion criteria Age 18 to 70 years Suspected PA admitted for diagnostic saline infusion testing or confirmed PA diagnosis according to Endocrine Society criteria.. Written informed consent

Exclusion criteria

* Age <18 or > 70 years.
* Pregnancy.
* Known adrenal failure and/or on steroid therapy (oral, inhaled, parenteral or topical) or other interfering medication.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected primary aldosteronism admitted to Haukeland University for diagnostic saline infusion test will be invited for study inclusion for dynamic microdialysis during saline infusion testing. If the diagnosis is confirmed, a repeated microdialysis sampling will be performed without saline infusion suppression.
  Additional patients with confirmed primary aldosteronism admitted to Haukeland University Hospital for subtyping with adrenal vein sampling will be invited for study inclusion for microdialysis without and during dexamethasone suppression.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Multisteroid rhythmicity of mineralocorticoids and glucocorticoids in primary aldosteronism | 2024-2028
  Assess multisteroid rhythmicity measured in microdialysis fluid of aldosterone, precursors and metabolites of the mineralocorticoid and glucocorticoid pathway, compared to standard diagnostic work-up in patients with suspected or confirmed PA.

SECONDARY OUTCOMES:
Effect of saline infusion test on multisteroid rhythmicity of mineralocorticoids and glucocorticoids | 2024-2028
  Influence of diagnostic saline infusion test on multisteroid adrenal rhythmicity will be assessed by performing 24h microdialysis before and during saling infusion testing
Effect of exogenous glucocorticoid suppression on aldosterone rhythmicity | 2024-2028
  Influence of exogenous administered glucocorticoids on aldosterone and related adrenal hormone rhythmicity will be assessed by performing 24h microdilays without and during suppression with exogenous glucocorticoids
cortisol co-secretion in primary aldosteronism | 2024-2028
  determine and quantify the presence of cortisol co-secretion in primary aldosteronism assessed by dynamic microdialysis compared with conventional cortisol co-secretion testing
Blood pressure, glucose and sleeep pattern correlation to dynamic hormone rhythmicity in primary aldosteronism | 2024-2028
  Correlate continous blood pressure and glucose variations, sleep, food intake and movement to variations in multisteroid hormone rhythmicity in primary aldosteronism.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Aarda Grytaas, MD PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided